CLINICAL TRIAL: NCT01906775
Title: Sub-threshold Ventricular Back-up Pacing to Prevent Pacemaker-induced Ventricular Tachycardia
Brief Title: Sub-threshold Pacing to Prevent Pacemaker-induced Ventricular Tachycardia
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Thomas Rostock, Univ.-Prof. Dr. med., Johannes Gutenberg University Mainz
Other Study IDs: PIT in ICD patients
Record Dates: First submitted 2013-07-20; First posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Ventricular Tachyarrhythmias; ICD Shock Therapy; ICD Shock Burden
Keywords: ICD; ventricular tachyarrhythmia; shock; sub-threshold pacing
MeSH Terms: conditions — Tachycardia, Ventricular; Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with PIT: Identification of patients with pacemaker-induced ventricular tachycardias
  Interventions: Other: Programming the pacemaker output for ventricular back-up pacing to a sub-threshold level

INTERVENTIONS:
Other: Programming the pacemaker output for ventricular back-up pacing to a sub-threshold level — Programming the pacemaker output for ventricular back-up pacing to a sub-threshold level to achieve an ineffective pacing output

SUMMARY:
Implantable cardioverter defibrillators (ICD) may have the capacity to provoke or worsen ventricular tachyarrhythmias (VT). It has been reported that ICD shocks by itself can increase mortality. This study aimed to determine the role of back-up pacing-induced VT (PIT) to the overall ICD shock burden by avoiding pause-related ventricular back-up pacing by programming the pacing output to a sub-threshold level for ineffective pacing.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* implanted ICD
* occurrence of pacemaker-induced VT

Exclusion Criteria:

* documentation of pause-related syncope
* AV block
* sick-sinus syndrome
* younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having an implanted ICD for secondary prevention of ventricular tachyarrhythmias. Patients are routinely under follow-up for device interrogation in our outpatient device department.
  Patients with identified pacemaker-induced ventricular tachycardia were selected and after two or more episodes of VT, the ventricular back-up pacing was reprogrammed to a sub-threshold level.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2003-06; Primary Completion 2012-09 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of VT requiring ICD shock | 48 months follow-up
  Patients were followed-up for the occurrence of ventricular tachycardia requiring ICD shock therapy

SECONDARY OUTCOMES:
Type of arrhythmia / Number of arrhythmia | 48 months
  Analysis of the number and the types of recurrent arrhythmias requiring ICD shock termination

OTHER OUTCOMES:
Incidence of PIT versus other VTs | 48 months
  Measurement of the proportion of PIT versus other VTs requiering ICD shock termination

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Mainz, II. Medical Clinic, Dept. of Electrophysiology, Mainz, Germany

REFERENCES:
- [Derived] Theis C, Mollnau H, Sonnenschein S, Konrad T, Himmrich E, Bock K, Schulz E, Kampfner D, Gerhardt S, Quesada Ocete B, Munzel T, Rostock T. Reduction of ICD shock burden by eliminating back-up pacing induced ventricular tachyarrhythmias. J Cardiovasc Electrophysiol. 2014 Aug;25(8):889-895. doi: 10.1111/jce.12418. Epub 2014 May 2. PMID 24654876